CLINICAL TRIAL: NCT00672815
Title: The Impact of Texas Senate Bill 42 on Middle School Children's Level of Physical Activity
Acronym: TXSB42
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Cristina S. Barroso, DrPH, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-SPH-06-0155; 56318 Active Living Research
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2010-01

CONDITIONS: Obesity; Body Weight
Keywords: coordinated school health; school health policy evaluation; physical activity
MeSH Terms: conditions — Obesity; Body Weight; Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study was twofold: 1) to assess awareness of and adherence to Texas SB42 among a representative sample of public middle schools in Texas; and 2) to assess the impact of SB42 on the frequency of school PE class, the quality of school PE, and prevalence of child self-reported physical activity behaviors and child overweight along the Texas-Mexico border.

DETAILED DESCRIPTION:
Childhood overweight is a significant public health issue in Texas. In response to this problem, the 79th Texas legislature passed Senate Bill 42 (SB 42), which promotes healthier school environments in middle schools, in June, 2005. As a result of SB 42, all Texas public middle schools must require students to engage in at least 30 minutes of daily physical activity or a total of 135 minutes of physical activity per week, beginning in the 2006-2007 school year. The purpose of this study was to determine the barriers and facilitators of implementation and the ultimate impact of this mandate on school PE, child physical activity, and child overweight in Texas public middle schools, and specifically among children living in the Lower Rio Grande Valley (LRGV) of South Texas. Questionnaires with key informants (school principals, PE teachers, and school district PE and health education directors) were conducted in a random sample of middle schools to assess the implementation of SB 42 (2006-2007). In addition, a more detailed evaluation of SB 42 was accomplished with a representative sample of middle schools in the LRGV, a low-income Latino area of the state. Measurements in the LRGV schools included observed and measured child physical activity, self-reported physical activity behaviors, and child overweight (BMI).

ELIGIBILITY:
Inclusion Criteria:

* The study sample consisted of a representative sample of Texas public middle schools (112 schools) as well as a representative sample of Lower Rio Grande Valley middle schools (17 schools).

Exclusion Criteria:

* Middle schools that did not participate in the 2004-2005 School Physical Activity and Nutrition Project.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are 1,224 school districts and 1,159 public middle schools in the state of Texas. Of all Texas students, 43% are Hispanic, 14% are African American, 40% are White, and 3% are other. Additionally, 51.8% are considered economically disadvantaged. PHR 11 covers a large area of the LRGV (along the Texas/Mexico border), and including 50 school districts and 485 public schools. Within PHR 11, 84.5% of children are considered economically disadvantage and more than 90% are Latino).
Sampling Method: Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
key informant questionnaire | April 2006- April 2008
System for Observing Fitness Instruction Time | April 2007 - April 2008
School Physical Activity Nutrition questionnaire | April 2007 - April 2008
body mass index | April 2007 - April 2008

CONTACTS AND LOCATIONS:
Overall Officials: Cristina S Barroso, DrPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center, Houston, Brownsville, Texas, United States

REFERENCES:
- [Result] Barroso CS, Kelder SH, Springer AE, Smith CL, Ranjit N, Ledingham C, Hoelscher DM. Senate Bill 42: implementation and impact on physical activity in middle schools. J Adolesc Health. 2009 Sep;45(3 Suppl):S82-90. doi: 10.1016/j.jadohealth.2009.06.017. PMID 19699442